CLINICAL TRIAL: NCT00873834
Title: Fluoxetine : Clinical and Anatomy-functional Therapeutic Effects in Children With Autism
Brief Title: Fluoxetine Essay in Children With Autism
Acronym: FAIR
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn for problem of logistics with the associated laboratories
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P030901; AOM 98082 (Other: French Ministry)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2009-04

CONDITIONS: Autism
Keywords: autism; fluoxetine; Comparative; double blind; placebo; controlled trial; anatomy-functional imaging; children; DSM-IV-R criteria for autism and CARS score (of 30 or above)
MeSH Terms: conditions — Autistic Disorder | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluoxetine arm (Experimental): Treatment with fluoxetine in an oral solution will be given at 0.25mg/kg day during 2 weeks and at 0.4mg/kg day during 16 weeks.
  A progressive decreased of dosage on a period of 4 weeks to 0.25mg/kg/day (2 weeks) and 0.10mg/kg/day(2 weeks) will be realized
  Interventions: Drug: fluoxetine
- placebo arm (Placebo Comparator): Placebo comparator. The packaging of study drug and placebo will be performed according to applicable regulatory requirements in the same packaging. An oral solution will be administrated.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: fluoxetine — Treatment with fluoxetine in an oral solution will be given at 0.25mg/kg day during 2 weeks and at 0.4mg/kg day during 16 weeks.
  A progressive decreased of dosage on a period of 4 weeks to 0.25mg/kg/day (2 weeks) and 0.10mg/kg/day(2 weeks) will be realized
  Other Names: SSRI compared to placebo
  Arms: Fluoxetine arm
Drug: placebo — Placebo comparator. The packaging of study drug and placebo will be performed according to applicable regulatory requirements in the same packaging. An oral solution will be administrated.
  Other Names: Placebo and drug packaging applied
  Arms: placebo arm

SUMMARY:
This study is a comparative, double blind, placebo controlled trial of 6-months duration designed to evaluate 1) the effects of fluoxetine in 5 to 12 years old autistic children, 2) the effects of fluoxetine on serotoninergic parameters, 3) cerebral metabolic changes (rCBF measurements with PET) induced by the treatment.

DETAILED DESCRIPTION:
Autism is a severe neurodevelopmental disorder characterized by impaired social interaction and communication, and by a markedly restricted repertoire of activities and interests. The population prevalence of autism is approximately 1 in 1000 (GILLBERG and WING, 1999) and the ratio of affected males to females is 4:1 (FOMBONNE, 1999). Although typically considered a childhood disorder, most persons with autism experience marked functional impairment throughout their lives. Follow-up studies of children with autism show that only 5%-10% become independent as adults, 25% progress but still require supervision, and the remaining continue to be severely impaired and in need of institutionalized care (WING, 1989). Thus, the syndrome represents a substantial public health problem with tragic cost to the individual, the family, and the community.

It is a randomized, double blind flexible dose study with parallel groups, controlled, fluoxetine versus placebo.

The final efficacy evaluation will be done after 6 months of treatment; Nine obligatory visits are planned Patients will be assessed at the following visits: base-line inclusion (D-15), and 2, 4, ,12, ,20, 22, 24 25, 26 weeks. At the 24 W visit, the final efficacy will be performed and medication will be tapered over a maximum period of 2 weeks. The final safety assessment will be performed at 26W.

BRAIN IMAGING PROTOCOL :

We will assess the resting state regional cerebral blood flow (rCBF) in autistic children using labeled water and PET, as it is still the most reliable and least invasive method. In addition, an anatomical and functional MRI will be performed in all children, the same day. Brain imaging studies will be performed at the Service HOSPITALIER Frederic JOLIOT (ORSAY, France) under Dr Monica ZILBOVICIUS responsibility.

Each brain imaging examination will be performed twice: 1) at time zero (T0) - before the beginning of the treatment and 2) six month later, after placebo or sertraline treatment.

Functional imaging in the resting state - Positron emission tomography :

Regional cerebral blood flow (rCBF) will be measured on a Siemens ECAT HR+ camera. Attenuation-corrected data are reconstructed into 63 slices, with a resulting resolution of 4.5 mm full-width-at-half-maximum. Fifteen seconds before each scan, 7 mCi of H215O is administrated by bolus injection. Data are collected during 80 s. All rCBF examinations will be performed at rest during sleep induced by premedication (4 mg/kg of pentobarbital). We have previously reported that this premedication has no effects on absolute rCBF values and regional distribution.

Anatomical MRI:

A high resolution MRI of the brain will be obtained in all children witg a 1.5 Tesla Signa General Electric scanner using a 3D T1-weighted FSPGR sequence (TR/TE/TI/NEX: 10.5/2.2/600/1, flip angle 10°, matrix size 256 x 192, yielding 124 axial slices and a thickness of 1.2 mm, field of view 22 cm). The acquisition duration is 6 minutes. In addition, FLAIR and T2 axial and coronal sequences will be also acquired.

Biological measures:

Blood sample procedure for whole blood serotonin: patients must follow a diet poor in tryptophan during two days before the blood sampling. Blood sample will be performed without premedication between nine and 11 AM. Blood will be withdrawn into tubes containing EDTA acid and aprotinin. Platelet- poor plasma (containing up to 0.1% of the original platelet count as assessed by contrast phase microscopy) is obtained within 2 hours by centrifugation (2000g, 4C, 15 mn) and frozen as 0.5mL aliquots at -80C until assess (blind procedures will be used). The whole blood content will by measured by radio-enzymology.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with diagnosis of Pervasive developmental disorder (PDD) meeting all criteria listed bellow will be included in the study:
* age 5 to 12 years, outpatients.
* presenting with a primary diagnosis of autism according to DSM- IV-R.
* Autism will be diagnosed with Autism Diagnostic Interview (ADI)
* with a score of 30 or above on the Children Autistic Rating Scale (CARS, SCHOPLER et al., 1980).
* Written informed consent obtained from each patient's parents or legal guardian.

Exclusion Criteria:

* Subjects presenting with any of the following will not be included in the study:
* Participation in any other studies involving investigational or marketed products within 6 months prior to entry in the study.
* Treatment given for autism within the previous 1 month
* Organic mental disorder or organic brain syndrome (including epilepsy)
* Severe mental retardation (IQ < 45).
* Specific systemic diseases, including history of significant hematological, endocrine, cardiovascular, renal, gastrointestinal or neurological disease (including more than one episode of childhood febrile convulsion).
* Medical contra-indication to treatment with any antidepressant and specially sertraline
* Previous history of intolerance or hypersensitivity to fluoxetine or to drugs with similar chemical structures
* Currant use of concomitant anticoagulant therapy
* Previous participation in any other clinical trial with the study drug
* Require concomitant therapy with any psychotropic drug or with any drug with a psychotropic component

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2010-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Subscores of Autism Diagnostic Interview (ADI-R)at each visit of the protocol (LECOUTER et RUTTER, 1989) | 6 months

SECONDARY OUTCOMES:
Sides effect scale (FSEC) | 6 months
Aberrant Behavior Checklist (Aman et al., 1985) | 6 months
Clinical Global Impressions (CGI) severity and improvement (NIMH.1985) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: CHABANE Nadia, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris (Hopital Robert DEBRE)